CLINICAL TRIAL: NCT02574286
Title: An Open-label, Multicenter, Single-arm, Phase 4 Study of the Effect of Treatment With Velaglucerase Alfa on Bone-related Pathology in Treatment-naïve Patients With Type 1 Gaucher Disease
Brief Title: Study of the Effect of Velaglucerase Alfa (VPRIV®) on Bone-related Pathology in Treatment-naïve Participants With Type 1 Gaucher Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP-GCB-402; 2015-001578-17 (EudraCT Number)
Record Dates: First submitted 2015-10-09; First posted 2015-10-12 (Estimated); Results first posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease | interventions — Glucosylceramidase; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Velaglucerase alfa 60 U/kg (Experimental): Participants will receive 60-minute intravenous infusion of 60 units per kilogram (U/kg) velaglucerase alfa every other week (EOW) and an oral daily dose of 800 IU vitamin D for 24 months (101 weeks).
  Interventions: Drug: Velaglucerase alfa; Dietary Supplement: Vitamin D

INTERVENTIONS:
Drug: Velaglucerase alfa — Participants will receive 60-minute intravenous infusion of 60 U/kg velaglucerase alfa EOW.
Dietary Supplement: Vitamin D — Participants will receive 800 IU vitamin D orally daily.

SUMMARY:
The primary purpose of this study is to evaluate the effect of VPRIV therapy (60 units per kilogram [U/kg] every other week [EOW]) in treatment-naive participants with type 1 Gaucher disease on change from baseline in lumbar spine (LS) bone mineral density (BMD) Z-score as measured by dual energy x-ray absorptiometry (DXA) after 24 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a documented diagnosis of type 1 Gaucher disease, as documented by deficient GCB activity in leukocytes (whole blood only) or cultured skin fibroblasts. Diagnosis by only dry blood spot test is insufficient. Diagnosis may be based on results obtained prior to screening if documented in the participant's medical history.
* Participants must have a LS BMD Z-score less than (<) -1 or BMD T-score of < -1 as measured by DXA during the screening phase.
* Participant is treatment-naive, that is (ie,) has not received ERT or SRT in the 12 months prior to enrollment.
* The participant is greater than or equal to (>=) 18 and less than or equal to (<=) 70 years of age.
* Female participants of childbearing potential must agree to use a medically acceptable method of contraception at all times during the study.
* The participant, or participant's legally authorized representative(s), if applicable, understands the nature, scope, and possible consequences of the study and has provided written informed consent that has been approved by the Institutional Review Board/Independent Ethics Committee (IRB/IEC).
* The participant must be sufficiently cooperative to participate in this clinical study as judged by the investigator.

Exclusion criteria

* Neurological symptoms indicating that the participant may have type 3 Gaucher disease.
* A significant comorbidity, which, as determined by the investigator, might affect study data or confound the study results (eg, malignancies, primary biliary cirrhosis, autoimmune liver disease, etc).
* Any osteoporosis-specific treatment (eg, bisphosphonates) or treatment with erythropoietin (or erythropoietin-like substances) during the past year.
* Structural, joint-associated bone damage of such extent and severity that the investigator deems it could impact participation in the study and assessment of relevant study endpoints (example, pain).
* The participant is pregnant or lactating.
* The participant has had a splenectomy. (This criterion is not meant to exclude participants who have accessory spleens.)
* The participant is enrolled in another clinical study that involves clinical investigations or use of any investigational product (drug or device) within 30 days prior to study enrollment or at any time during the study.
* Severe vitamin D deficiency to the level that would be expected to result in osteomalacia (vitamin D < 10 nanograms per milliliter [ng/mL] [25 nanomoles per liter {nmol/L}]). If there is mild vitamin D insufficiency at screening (vitamin D greater than [>] 10 and < 30 ng/mL) treat with 4000 IU vitamin D per day for 1 month and rescreen.
* The participant has previously interrupted ERT for safety reasons.
* The participant has had hypersensitivity to the active substance or to any of the excipients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (15):
- United States (8):
  - Cedars Sinai Medical Center, Beverly Hills, California
  - Kaiser Permanente, Los Angeles, California
  - Emory Genetics, Atlanta, Georgia
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - NYU School of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Lysosomal and Rare Disorders Research and Treatment Center, Fairfax, Virginia
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
- Spain (2):
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Quironsalud Zaragoza, Zaragoza
- United Kingdom (2):
  - Addenbrooke's Hospital, Cambridge
  - Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in the United States, Israel, Spain and United Kingdom from 29 June 2016 (first participants first visit) to 30 November 2020 (last participants last visit).
Pre-assignment Details: A total of 21 participants were enrolled and received treatment in this study.
Groups:
- Velaglucerase Alfa 60 U/kg: Participants received 60-minute intravenous (IV) infusion of 60 units per kilogram (U/kg) velaglucerase alfa every other Week (EOW) for 24 months (up to 101 weeks).
Period: Overall Study
Arm/Group | Velaglucerase Alfa 60 U/kg
Started | 21
Completed | 16
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Safety population was defined as all enrolled participants who received at least one study drug infusion (full or partial).
Groups:
- Velaglucerase Alfa 60 U/kg: Participants received 60-minute intravenous (IV) infusion of 60 units per kilogram (U/kg) velaglucerase alfa EOW for 24 months (up to 101 weeks).
Arm/Group | Velaglucerase Alfa 60 U/kg
Number analyzed (Participants) | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 1
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.9 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Lumbar Spine Bone Mineral Density (BMD) Z-Score up to End of Study (EOS) (Week 103)
Description: Bone mineral density of the lumbar spine was measured by dual energy x-ray absorptiometry (DXA), and the results was converted to Z-scores appropriate for age, sex, and race. The Z-score indicated the number of standard deviations away from a reference population in the same age range, race and with the same sex. A Z-score of 0 was equal to the mean. Negative numbers indicated values lower than the mean and positive numbers indicated values higher than the mean. Baseline was defined as last data collected prior to the first administration of study drug. Change from baseline in lumbar spine BMD Z-Score up to EOS (Week 103) was reported.
Time Frame: Baseline up to EOS (Week 103)
Population: Intent-to-Treat (ITT) Population was defined as all enrolled participants who received at least one study drug infusion (full or partial). Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Velaglucerase Alfa 60 U/kg
Number analyzed (Participants) | 16
Z-score | 0.17 (0.394)

2. Secondary Outcome: Change From Baseline in Lumbar Spine (LS) BMD Z-score at Week 51
Description: BMD of the LS was measured by DXA, and the results was converted to Z-scores appropriate for age, sex, and race. The Z-score indicated the number of standard deviations away from a reference population in the same age range, race and with the same sex. A Z-score of 0 was equal to the mean. Negative numbers indicated values lower than the mean and positive numbers indicated values higher than the mean. Baseline was defined as last data collected prior to the first administration of study drug. Change From baseline in LS BMD Z-score at Week 51 was reported. ITT Population was defined as all enrolled subjects who received at least one study drug infusion (full or partial). Here, "number of subjects analysed" signifies subjects who were evaluable for this endpoint.
Time Frame: Baseline, Week 51
Population: ITT Population was defined as all enrolled participants who received at least one study drug infusion (full or partial). Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Velaglucerase Alfa 60 U/kg
Number analyzed (Participants) | 16
Z-Score | 0.02 (0.431)

3. Secondary Outcome: Change From Baseline in Lumbar Spine BMD at Week 51 and EOS (Week 103)
Description: Bone mineral density of the LS was measured by DXA, and the results was measured in gram per square centimeter (g/cm^2). Baseline was defined as last data collected prior to the first administration of study drug. Change From baseline in LS BMD at Week 51 and EOS (Week 103) was reported.
Time Frame: Baseline, Week 51 and EOS (Week 103)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Velaglucerase Alfa 60 U/kg
Number analyzed (Participants) | 16
g/cm^2
  Change at Week 51 | 0.006 (0.0342)
  Change at EOS (Week 103) | 0.011 (0.0474)

4. Secondary Outcome: Change From Baseline in Total Bone Marrow Burden (BMB) Score at Week 51 and EOS (Week 103)
Description: BMB score was a semi-quantitative magnetic resonance imaging (MRI) scoring system for assessing the extent of bone marrow involvement in Gaucher disease. BMB Score was measured using magnetic resonance imaging (MRI), range from 0 (no abnormalities) to 8 points (severe disease) for the lumbar spine and from 0 (no abnormalities) to 8 points (severe disease) for the femurs. The total BMB score was calculated as the sum of scores for femur and lumbar spine regions which ranged from 0 (no abnormalities) to 16 (severe disease) points. A higher BMB score signified more severe bone marrow involvement. Baseline was defined as last data collected prior to the first administration of study drug. Change from baseline in total BMB Score at Week 51 and EOS (Week 103) was reported.
Time Frame: Baseline, Week 51 and EOS (Week 103)
Population: ITT Population was defined as all enrolled participants who received at least one study drug infusion (full or partial). Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants evaluable at specific time point.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Velaglucerase Alfa 60 U/kg
Number analyzed (Participants) | 15
Score on a Scale
  Change at Week 51 | -3.0 (1.85)
  Change at EOS (Week 103): number analyzed (Participants) | 13
  Change at EOS (Week 103) | -3.0 (2.27)

5. Secondary Outcome: Change From Baseline in Hemoglobin Concentration at Week 13, 25, 37, 51, 65, 77, 89, and EOS (Week 103)
Description: Blood samples were collected for measurement of hemoglobin concentration. Baseline was defined as last data collected prior to the first administration of study drug. Change from baseline in hemoglobin concentration at Week 13, 25, 37, 51, 65, 77, 89, and EOS (Week 103) was reported.
Time Frame: Baseline, Week 13, 25, 37, 51, 65, 77, 89, and EOS (Week 103)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Grams per deciliter (g/dL)
Arm/Group | Velaglucerase Alfa 60 U/kg
Number analyzed (Participants) | 18
Grams per deciliter (g/dL)
  Change at Week 13: number analyzed (Participants) | 17
  Change at Week 13 | 0.532 (0.7624)
  Change at Week 25 | 0.764 (0.6688)
  Change at Week 37: number analyzed (Participants) | 17
  Change at Week 37 | 0.765 (0.7836)
  Change at Week 51: number analyzed (Participants) | 17
  Change at Week 51 | 0.935 (0.6588)
  Change at Week 65: number analyzed (Participants) | 17
  Change at Week 65 | 1.029 (0.8239)
  Change at Week 77: number analyzed (Participants) | 13
  Change at Week 77 | 1.015 (1.1577)
  Change at Week 89: number analyzed (Participants) | 13
  Change at Week 89 | 1.138 (0.8910)
  Change at Week EOS (Week 103) | 0.897 (1.2309)

6. Secondary Outcome: Change From Baseline in Platelet Count at Week 13, 25, 37, 51, 65, 77, 89, and EOS (Week 103)
Description: Blood samples were collected for measurement of platelet count. Baseline was defined as last data collected prior to the first administration of study drug. Change from baseline over time in platelet count at Week 13, 25, 37, 51, 65, 77, 89, and EOS (Week 103) was reported.
Time Frame: Baseline, Week 13, 25, 37, 51, 65, 77, 89, and EOS (Week 103)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: 10^9 platelets per liter
Arm/Group | Velaglucerase Alfa 60 U/kg
Number analyzed (Participants) | 17
10^9 platelets per liter
  Change at Week 13: number analyzed (Participants) | 16
  Change at Week 13 | 38.06 (35.571)
  Change at Week 25 | 53.24 (46.955)
  Change at Week 37: number analyzed (Participants) | 15
  Change at Week 37 | 62.23 (46.834)
  Change at Week 51: number analyzed (Participants) | 16
  Change at Week 51 | 79.66 (89.701)
  Change at Week 65: number analyzed (Participants) | 16
  Change at Week 65 | 75.03 (52.163)
  Change at Week 77: number analyzed (Participants) | 13
  Change at Week 77 | 87.19 (70.528)
  Change at Week 89: number analyzed (Participants) | 12
  Change at Week 89 | 71.96 (60.772)
  Change at EOS (Week 103): number analyzed (Participants) | 16
  Change at EOS (Week 103) | 69.16 (53.451)

7. Secondary Outcome: Change From Baseline in Normalized Liver Volume at Week 51 and EOS (Week 103)
Description: Normalized liver volume was measured by abdominal MRI. Baseline was defined as last data collected prior to the first administration of study drug. Liver volume has been normalized for percent (%) body weight. Liver size relative to body weight = (Liver volume [cubic centimeter (cc)]/Body weight [kg])*100. Change from baseline in normalized liver volume at Week 51 and EOS (Week 103) was reported.
Time Frame: Baseline, Week 51 and EOS (Week 103)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent body weight
Arm/Group | Velaglucerase Alfa 60 U/kg
Number analyzed (Participants) | 17
Percent body weight
  Change at Week 51 | -0.353 (0.3485)
  Change at EOS (Week 103): number analyzed (Participants) | 15
  Change at EOS (Week 103) | -0.447 (0.4048)

8. Secondary Outcome: Change From Baseline in Normalized Spleen Volume at Week 51 and EOS (Week 103)
Description: Normalized spleen volume was measured by MRI. Spleen volume was normalized for % of body weight. Spleen size relative to body weight= (Spleen volume [cc]/Body weight [kg])*100. Baseline was defined as last data collected prior to the first administration of study drug. Change from baseline in normalized spleen volume at Week 51 and EOS (Week 103) was reported.
Time Frame: Baseline, Week 51 and EOS (Week 103)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent body weight
Arm/Group | Velaglucerase Alfa 60 U/kg
Number analyzed (Participants) | 17
Percent body weight
  Change at Week 51 | -0.443 (0.5987)
  Change at EOS (Week 103): number analyzed (Participants) | 15
  Change at EOS (Week 103) | -0.556 (0.7398)

9. Secondary Outcome: Change From Baseline in Severity of Bone Pain at Week 51 and EOS (Week 103)
Description: Bone pain was measured by questions taken from the Brief Pain Inventory-short form (BPI-SF). Pain severity was evaluated based on the average of 4 questions from BPI-SF (Questions 3 through 6) assessing worst pain, least pain, average pain, and pain right now, each rated on a scale from 0 (no pain) to 10 (pain as bad as you can imagine) with mild pain- score (1 to 4), moderate pain- score (5 to 6), and severe pain score (7 to 10). Overall severity score was calculated as average of 4 questions ranging from 0 (no pain) to 10 (pain as bad as you can imagine). A negative change from baseline score indicates improvement. Baseline was defined as last data collected prior to the first administration of study drug. Change from baseline in severity of bone pain at Week 51 and EOS (Week 103) was reported.
Time Frame: Baseline, Week 51 and EOS (Week 103)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Velaglucerase Alfa 60 U/kg
Number analyzed (Participants) | 1
Score on a Scale
  Change at Week 51 | -2.750 (NA) — Here "NA" signifies standard deviation was not estimated due to single participant.
  Change at EOS (Week 103) | -3.250 (NA) — Here "NA" signifies standard deviation was not estimated due to single participant.

10. Secondary Outcome: Change From Baseline in Bone Pain Interference Score at Week 51 and EOS (Week 103)
Description: Bone pain interference was measured by questions taken from the BPI-SF. Pain interference was evaluated based upon average of 7 questions from BPI-SF (9A through 9G) regarding the extent to which pain interfered with daily activities, including general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life in the last 24 hours, each rated on a scale from 0 (does not interfere) to 10 (completely interferes). Overall pain interference score was calculated as average of 7 questions ranging from 0 (does not interfere) to 10 (completely interferes). A negative change from baseline score indicates improvement. Baseline was defined as last data collected prior to the first administration of study drug. Change from baseline in bone pain interference score at Week 51 and EOS (Week 103) was reported.
Time Frame: Baseline, Week 51 and EOS (Week 103)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Velaglucerase Alfa 60 U/kg
Number analyzed (Participants) | 1
Score on a Scale
  Change at Week 51 | -1.286 (NA) — Here "NA" signifies standard deviation was not estimated due to single participant.
  Change at EOS (Week 103) | -4.429 (NA) — Here "NA" signifies standard deviation was not estimated due to single participant.

11. Secondary Outcome: Change From Baseline in Overall Fatigue Measured by Brief Fatigue Inventory (BFI) at Week 51 and EOS (Week 103)
Description: Overall fatigue was measured by the BFI. BFI was a 9-item questionnaire developed to assess subjective fatigue. Each question asked the respondent to rate the level of their experienced fatigue over the past 24 hours on an 11-point (0-10) scale. First 3 questions measure fatigue severity at current, usual, and worst levels, respectively, with 0 indicating "no fatigue" and 10 indicating fatigue "as bad as you can imagine". Next 6 questions assessed the level fatigue interference with daily activities included general activity, mood, walking ability, normal work (both inside and outside the home), relations with other people, and enjoyment of life. A score of 0="no interference" while a score of 10="complete interference. Overall fatigue score was calculated as average score of all 9 items on the BFI ranging from 0="no fatigue" to 10="as bad as you can imagine".
Time Frame: Baseline, Week 51 and EOS (Week 103)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Velaglucerase Alfa 60 U/kg
Number analyzed (Participants) | 5
Score on a Scale
  Change at Week 51 | -0.111 (1.4551)
  Change at EOS (Week 103) | 0.044 (3.7132)

12. Secondary Outcome: Number of Participants With Shift in World Health Organization (WHO) BMD Classifications Based on LS T-Scores at Week 51 and EOS (Week 103)
Description: WHO BMD Classifications (Normal Bone Density, Osteopenia, Osteoporosis), bone mineral density was classified based on LS BMD T-scores. BMD T-score was a comparison of an individual's BMD compared to "normal". Also, BMD T-score is the standard deviation of the difference between measured BMD and that of the healthy young adult "normal". The T-score scale was as follows: -1 and above=normal, -1 to -2.5=osteopenia (below normal and may lead to osteoporosis), and -2.5 and below=osteoporosis. Number of participants with shift in WHO BMD classifications based on LS T-Scores at Week 51 and EOS (Week 103) were reported.
Time Frame: Baseline, Week 51 and EOS (Week 103)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Velaglucerase Alfa 60 U/kg
Number analyzed (Participants) | 16
Participants
  Normal at Baseline- Normal at Week 51: number analyzed (Participants) | 0
  Normal at Baseline- Normal at Week 51 | 0
  Normal at Baseline- Osteopenia at Week 51: number analyzed (Participants) | 0
  Normal at Baseline- Osteopenia at Week 51 | 0
  Normal at Baseline- Osteoporosis at Week 51: number analyzed (Participants) | 0
  Normal at Baseline- Osteoporosis at Week 51 | 0
  Osteopenia at Baseline- Normal at Week 51: number analyzed (Participants) | 10
  Osteopenia at Baseline- Normal at Week 51 | 1
  Osteopenia at Baseline- Osteopenia at Week 51: number analyzed (Participants) | 10
  Osteopenia at Baseline- Osteopenia at Week 51 | 6
  Osteopenia at Baseline- Osteoporosis at Week 51: number analyzed (Participants) | 10
  Osteopenia at Baseline- Osteoporosis at Week 51 | 3
  Osteoporosis at Baseline- Normal at Week 51: number analyzed (Participants) | 6
  Osteoporosis at Baseline- Normal at Week 51 | 0
  Osteoporosis at Baseline- Osteopenia at Week 51: number analyzed (Participants) | 6
  Osteoporosis at Baseline- Osteopenia at Week 51 | 0
  Osteoporosis at Baseline- Osteoporosis at Week 51: number analyzed (Participants) | 6
  Osteoporosis at Baseline- Osteoporosis at Week 51 | 6
  Normal at Baseline- Normal at Week 103: number analyzed (Participants) | 1
  Normal at Baseline- Normal at Week 103 | 1
  Normal at Baseline- Osteopenia at Week 103: number analyzed (Participants) | 1
  Normal at Baseline- Osteopenia at Week 103 | 0
  Normal at Baseline- Osteoporosis at Week 103: number analyzed (Participants) | 1
  Normal at Baseline- Osteoporosis at Week 103 | 0
  Osteopenia at Baseline- Normal at Week 103: number analyzed (Participants) | 10
  Osteopenia at Baseline- Normal at Week 103 | 2
  Osteopenia at Baseline- Osteopenia at Week 103: number analyzed (Participants) | 10
  Osteopenia at Baseline- Osteopenia at Week 103 | 6
  Osteopenia at Baseline- Osteoporosis at Week 103: number analyzed (Participants) | 10
  Osteopenia at Baseline- Osteoporosis at Week 103 | 2
  Osteoporosis at Baseline- Normal at Week 103: number analyzed (Participants) | 5
  Osteoporosis at Baseline- Normal at Week 103 | 0
  Osteoporosis at Baseline- Osteopenia at Week 103: number analyzed (Participants) | 5
  Osteoporosis at Baseline- Osteopenia at Week 103 | 0
  Osteoporosis at Baseline- Osteoporosis at Week 103: number analyzed (Participants) | 5
  Osteoporosis at Baseline- Osteoporosis at Week 103 | 5

13. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. A TEAE was defined as any AE that occurred on or after the time of the first infusion of study drug until 30 days after the last infusion of study drug. Number of participants with TEAEs were reported.
Time Frame: From start of study drug infusion up to follow-up (107 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Velaglucerase Alfa 60 U/kg
Number analyzed (Participants) | 21
Participants | 21

14. Secondary Outcome: Number of Participants Who Developed Positive Anti-velaglucerase Alfa Antibody Status
Description: Anti-velaglucerase alfa antibody included anti-velaglucerase antibodies (ADA) and neutralizing anti-velaglucerase antibodies (NAb). The Anti-velaglucerase antibody status was summarized as categorical variable by positive and negative. Number of participants who developed positive anti-velaglucerase alfa antibody were reported.
Time Frame: Baseline up to EOS (Week 103)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Velaglucerase Alfa 60 U/kg
Number analyzed (Participants) | 21
Participants | 1

ADVERSE EVENTS:
Time Frame: From start of study drug infusion up to follow-up (107 weeks)
Groups:
- Velaglucerase Alfa 60 U/kg: Subjects received 60-minute intravenous (IV) infusion of 60 units per kilogram (U/kg) velaglucerase alfa every other Week (EOW) for 24 months (up to 101 weeks).
Arm/Group | Velaglucerase Alfa 60 U/kg
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 2/21
Other Adverse Events (participants affected / at risk) | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Velaglucerase Alfa 60 U/kg (N=21)
Pyelonephritis (Infections and infestations) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Velaglucerase Alfa 60 U/kg (N=21)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (20)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (4)
Headache (Nervous system disorders) | 6 (15)
Dizziness (Nervous system disorders) | 5 (11)
Fatigue (General disorders) | 5 (6)
Asthenia (General disorders) | 3 (3)
Influenza like illness (General disorders) | 2 (2)
Injection site bruising (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (11)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasopharyngitis (Infections and infestations) | 5 (6)
Pneumonia (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (4)
Blood iron decreased (Investigations) | 2 (2)
C-reactive protein increased (Investigations) | 2 (2)
Eye pain (Eye disorders) | 3 (3)
Vitamin D deficiency (Metabolism and nutrition disorders) | 4 (4)
Depression (Psychiatric disorders) | 2 (2)
Bundle branch block right (Cardiac disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (4)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/86/NCT02574286/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/86/NCT02574286/SAP_001.pdf